CLINICAL TRIAL: NCT05175326
Title: Study on the Consistency Evaluation of Organoids Used in the Clinical Treatment of Ovarian Cancer With Anti-tumor Drugs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-294
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Cancer; Organoid
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, observational clinical study that plans to recruit 64 ovarian cancer patients within one year. The purpose of this study is to evaluate the consistency and accuracy of the organoid model derived from patients with ovarian cancer and the patient's clinical medication, so as to predict the clinical efficacy of anti-cancer drugs

ELIGIBILITY:
Inclusion Criteria:

- Patients with ovarian cancer who are diagnosed as ovarian cancer by tissue and/or cytology and need neoadjuvant, adjuvant or standard treatment Age 18-75 years old (including 18 years old and 75 years old) It is clear that there are measurable lesions (according to RECIST1.1)

Exclusion Criteria:

- Patients with concurrent radiotherapy and chemotherapy, less than half a year of radiotherapy, or patients undergoing radiotherapy during the study period During the study period, patients need other tumor treatment methods such as surgery, intervention, radiofrequency ablation, etc.

Immune deficiency or severe bone marrow suppression The patient has severe liver and kidney disease, cardiovascular disease, blood disease, etc.

Illegal use of drugs or chronic alcohol abuse or total daily alcohol intake> 50 g/d Lack of autonomy, unable to walk, or unable to participate in the 6-month follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histologically confirmed ovarian cancer from Sun Yat-sen Memorial Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of the response to treatment by the patient-derived organoids | 2021-2022
  The drug sensitivity was tested on patient-derived tumour organoids, which is compared with clinical response of the chemo- or targeted therapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rao Qunxian, Study Director — The Sun Yat-sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- The Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No